CLINICAL TRIAL: NCT05934019
Title: Randomized Controlled Trial on the Efficacy of a Transdiagnostic Online Prevention Approach in Adolescents (EMPATIA)
Brief Title: Efficacy of a Transdiagnostic Online Prevention Approach in Adolescents (EMPATIA)
Acronym: EMPATIA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-D0036
Record Dates: First submitted 2023-05-26; First posted 2023-07-06 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Mental Health Issue; Transdiagnostic Mechanisms; Adolescent Psychology; Prevention; Online Intervention; Psychological Intervention; Mental Disorder in Adolescence, Subclinical

STUDY DESIGN:
Intervention Model Description: The present study is a monocentric, two-arm, single-blinded, randomized controlled trial with CAU as control condition.
Who Masked: Outcomes Assessor
Masking Description: Study participants cannot be blinded regarding the intervention condition as they realize whether they are in the condition using an online-program or not. Members of the study team guiding the participants as e-coaches during the online-program cannot be blinded as it is obvious for them that this is the condition receiving the online-program. Members of the study team who are conducting the diagnostic interviews do not have any other contact with the participants and will thus be blinded regarding the participants' assignment to the group conditions (EMPATIA vs. CAU).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMPATIA (Experimental): Participants in this group will access the online prevention program EMPATIA as a self-help online program during eight weeks.
  Interventions: Device: EMPATIA 1
- Care As Usual (No Intervention): Participants in this group will gain access to the online prevention program EMPATIA after 12 months. All other kinds of interventions during participation are allowed and will be recorded using the Client Sociodemographic and Service Receipt Inventory

INTERVENTIONS:
Device: EMPATIA 1 — The internet-program EMPATIA is hosted on a secure website https://selfhelp.psy.unibe.ch run by the Faculty of Human Sciences and is accessible from any regular internet browser. The software is not CE-marked as it has been developed for research purposes only. EMPATIA consists of 8 sessions and 1 booster session 3 weeks after the last session. It targets transdiagnostic mechanisms that have been identified in several mental disorders in adolescents: behavioral avoidance, repetitive negative thinking including intolerance of uncertainty, emotion, self-critical perfectionism and rejection sensitivity. The contents of EMPATIA are evidence-based and well-established cognitive-behavioral interventions dedicated to the respective transdiagnostic mechanism. The self-help program consists of psychoeducation, cognitive restructuring, relaxation and acceptance-based interventions, exposure and behavioral experiments and behavioral activation as treatment components.
  Arms: EMPATIA

SUMMARY:
The goal of this randomized controlled clinical trial is to investigate the efficacy of the internet-delivered intervention EMPATIA on general psychopathology of adolescents with subclinical symptoms compared to a Care As Usual (CAU) control group. The primary objective is to:

* investigate the efficacy of the internet-delivered intervention on general psychopathology of adolescents with subclinical symptoms compared to CAU.
* secondary objectives include: clinician-rated interviews and self-report questionnaires on the level of social and role functioning, time until onset of a mental disorder and service use. Furthermore, changes in subclinical symptoms, transdiagnostic mechanisms and therapeutic as well as safety measures are assessed by online self-reports

Participants will use the internet-delivered intervention EMPATIA during eight weeks.

Researchers will compare intervention group to a Care As Usual (CAU) group to investigate the efficacy of the internet-delivered intervention EMPATIA on general psychopathology.

DETAILED DESCRIPTION:
The overall objective of this study is to develop and evaluate an internet-delivered indicated prevention program for adolescents with subclinical symptoms designed to target transdiagnostic mechanisms of change. The internet-delivered program will be evaluated in a RCT compared to Care As Usual (CAU) including a 1-year follow-up period.

The online program EMPATIA aims to strengthen the well-being and mental health of young people in the long term. For example, in this program, young people learn, among other things, how to better deal with worries, stress, low self-confidence, conflicts with other people, or even unpleasant feelings such as anger, fear, or sadness. These are skills that are known to be helpful for the further development of all adolescents and make them more resilient to stress.

In this study, the investigators want to investigate whether the program is helpful, how it works, and which adolescents profit most. For the study, 152 adolescents from Switzerland are asked to participate in the EMPATIA-program online. In order to study the effectiveness scientifically, all adolescents will be randomly divided into two groups, so the differences can be compared. One group will get access to the EMPATIA-program already at the beginning, the other group after 12 months.

The contents of the EMPATIA-Program are evidence-based and well-established cognitive-behavioural interventions targeting transdiagnostic mechanisms that have been repeatedly identified to underlie several mental disorders in adolescents: behavioral avoidance, repetitive negative thinking including rumination, worry and intolerance of uncertainty, emotion regulation, self-critical perfectionism and rejection sensitivity. The program consists of 8 modules. It is recommended to complete one module every week with each module lasting about 60 minutes and to make use of additional examples, exercises for everyday life and diaries as often as possible. Furthermore, age- and gender specific topics and main testimonials are offered and can be selected by each participant. The intervention allows tailoring contents through topics that can be additionally selected, such as interpersonal conflicts, self-esteem, and social support and additional examples (e.g., if the predominant emotion experienced is anger vs. sadness). Information will generally be presented via short video-clips, examples from testimonials, audio files, interactive elements, and cartoons instead of text-based parts. At the end of the modules, there is a short quiz that allows participants to review and solidify what they have learned.

Participants will be guided (via program integrated chat function) throughout the intervention by e-coaches who are advanced master-students in Clinical Child and Adolescent Psychology.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject (if the participant is ≥ 14 years) or signed by the legal guardians (if the participant is 12 or 13 years old).
* Subjects are between 12 and 18 years old.
* Subjects experience at least mild self-reported symptoms by scoring above the cut-off in at least one of the respective screening-instruments as assessed at the 12-month follow-up of the EMERGE- study.
* Subjects have access to the internet and a smart phone, tablet or personal computer.
* Subjects have sufficient knowledge of German.

Exclusion Criteria:

* Current or lifetime diagnosis according to the "Diagnostic Interview for Mental Disorders for Children and Adolescents" (Kinder-DIPS, Margraf et al., 2017; Schneider et al., 2017) at baseline.
* Score of '3' on the suicide item of the PHQ-A (Johnson et al., 2002) or active suicidal plans in the diagnostic telephone interview (Kinder- DIPS, Margraf et al., 2017; Schneider et al., 2017) at baseline.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Level of self-reported general psychopathology | Baseline
  Assessed by the "Strength and Difficulties Questionnaire, self-report" (SDQ-s; Becker et al., 2018). 25 Items with higher scores indicating higher level of self-reported general psychopathology.
Level of self-reported general psychopathology | Month 2
  Assessed by the "Strength and Difficulties Questionnaire, self-report" (SDQ-s; Becker et al., 2018). 25 Items with higher scores indicating higher level of self-reported general psychopathology.
Level of self-reported general psychopathology | Month 6
  Assessed by the "Strength and Difficulties Questionnaire, self-report" (SDQ-s; Becker et al., 2018). 25 Items with higher scores indicating higher level of self-reported general psychopathology.
Level of self-reported general psychopathology | Month 9
  Assessed by the "Strength and Difficulties Questionnaire, self-report" (SDQ-s; Becker et al., 2018). 25 Items with higher scores indicating higher level of self-reported general psychopathology.
Level of self-reported general psychopathology | Month 12
  Assessed by the "Strength and Difficulties Questionnaire, self-report" (SDQ-s; Becker et al., 2018). 25 Items with higher scores indicating higher level of self-reported general psychopathology.

SECONDARY OUTCOMES:
Level of social functioning | Baseline and month 12
  Assessed with a structured interview ("Global Functioning Social"; GFsocial; Cornblatt et al., 2007). Scores range from 1 to 10 with higher scores indicating higher social functioning.
Level of role functioning | Baseline and month 12
  Assessed with a structured interview ("Global Functioning Role"; GFrole; Cornblatt et al., 2007). Scores range from 1 to 10 with higher scores indicating higher role functioning.
Time until onset of a mental disorder | Baseline and month 12
  Assessed with the Kinder-DIPS ("Diagnostic Interview for Mental Disorders in Children and Adolescents"; Schneider, Pflug, In-Albon, & Margraf, 2017)
Service Use | Month 12
  Assessed with the German version of the "Client Sociodemographic and Service Receipt Inventory" (CSSRI-EU; Chisholm et al., 2000; Roick et al., 2001).
Depression | Baseline, Month 2, 6, 9 and 12
  The "Patient Health Questionnaire-9 for Adolescents" (PHQ-A; Johnson et al., 2002) will be used to assess depressive symptoms. This self-report questionnaire consists of 9 items and higher scores indicate higher depressive symptoms.
Hypomania/bipolar symptoms (ASRM; Altman et al., 1997) | Baseline, Month 2, 6, 9 and 12
  The "Altman Self-Rating Mania" Scale (ASRM) will be used to assess hypomania/bipolar symptoms. It is a 5-item Likert scale in which manic symptoms, corresponding to diagnostic criteria for mania, are rated from 0 to 4 according to increasing severity.
Anxiety (GAD-7; Löwe et al., 2008) | Baseline, Month 2, 6, 9 and 12
  The GAD-7 will be used to measure general anxiety symptoms with 7 items. Higher scores indicate higher levels of anxiety.
Obsessive-compulsive symptoms (SOCS; Piqueras et al., 2015) | Baseline, Month 2, 6, 9 and 12
  The "Short Obsessive-Compulsive Disorder Screener" (SOCS), a 6 item screening instrument, will be used to assess obsessive-compulsive symptoms.
Psychotic-like experiences (CAPE-P15; Capra et al., 2013). | Baseline, Month 2, 6, 9 and 12
  The 15 item self-report questionnaire CAPE-P15 (Capra et al., 2013) assesses three domains: paranoid ideation, bizarre experiences, and perceptual anomalies. Scores can range from 15 to 75. Higher scores indicate higher severity of psychotic-like experiences.
Alcohol/Substance abuse (CRAFFTd; Tossman et al., 2009) | Baseline, Month 2, 6, 9 and 12
  The CRAFFTd (Tossman et al., 2009) is a one-dimensional screening tool consisting of 6 questions. It will be used to screen for problematic substance consumption in adolescents. Higher scores indicate greater problematic substance consumption.
Eating behavior (ChEDE-Q8; Kliem et al., 2016) | Baseline, Month 2, 6, 9 and 12
  The "Child Eating Disorder Examination-Questionnaire" (ChEDE-Q8) used in this study is an 8 item self-report scale to assess specific eating disorder psychopathology.
Conduct disorder (SDQ-s; Becker et al., 2018) | Baseline, Month 2, 6, 9 and 12
  The subscale of the "Strengths and Difficulties Questionnaire" (SDQ-s; Becker et al., 2018) will be used to assess subclinical conduct problems. 5 items, higher scores indicate higher severity of conduct problems.
Non-suicidal self-injurious behavior | Baseline, Month 2, 6, 9 and 12
  (Kinder-DIPS, Additional-Module NSSV; Margraf et al., 2017; Schneider et al., 2017). The suggested 7 questions by Margraf et al. (2017) and Schneider et al. (2017) will be assessed via self-report. Non-suicidal self-injurious behavior in the past year on five or more separate occasions are considered as subclinical.
Somatic symptoms (SSS8; Gierk et al., 2014) | Baseline, Month 2, 6, 9 and 12
  The "Somatic Symptom Scale" (SSS-8) with 8-item will be used for the assessment of somatic symptom burden. Higher scores indicate higher somatic symptom burden.
Current stress level (PSS-4; Herrero & Meneses, 2006) | Baseline, Month 2, 6, 9 and 12
  "Perceived Stress Scale" to assess current levels of stress (PSS-4), 4-item version with responses scored on a 1- to 5-point scale.
Adjustment to daily life (WSAS-Y; Jassi et al., 2020) | Baseline, Month 2, 6, 9 and 12
  The WSAS-Y ("Work and Social Adjustment Scale-Youth") consists of five items that are rated on a 9-point Likert scale, generating a global score ranging from 0 to 40 (Jassi et al., 2020).
Behavioral avoidance (CEASE-A; Fairholm & Ehrenreich, 2008) | Baseline, Month 2, 6, 9 and 12
  The "Checklist of Avoidance Strategy Engagement for Adolescents" (CEASE-A) is a psychometrically sound measure of avoidance (Kennedy, 2015). The 29-item checklist assesses frequency of engagement in avoidance behaviors to manage or avoid feelings of anxiety, anger, fear, or sadness on a 5-point Likert-type scale.
Self-perfectionism (F-MPS-B; Burgess et al., 2016) | Baseline, Month 2, 6, 9 and 12
  The "Frost Multi-Dimensional Perfectionism Scale-Brief" (F-MPS-B; Burgess et al. 2016) is a brief 8-item version of the original F-MPS (35-items) (Frost et al. 1990). Items are rated on a 5-point Likert type scale with higher scores indicating greater perfectionism.
Repetitive negative thinking (RTQ-10; McEvoy et al., 2017) | Baseline, Month 2, 6, 9 and 12
  The "Repetitive Thinking Questionnaire" (RTQ-10) is a 10-item scale to measure the common transdiagnostic factor repetitive negative thinking. Items are rated on a 5-point scale.
Emotion regulation (DERS-16; Bjureberg et al., 2016) | Baseline, Month 2, 6, 9 and 12
  The "Difficulties in Emotion Regulation Scale" (DERS-16) is a 16-item self- report measure of emotion regulation difficulties (Bjureberg et al., 2016).
Intolerance of Uncertainty (IUS-12; Carleton et al., 2012) | Baseline, Month 2, 6, 9 and 12
  The "Intolerance of Uncertainty Scale" is a 12-item short-form of the original 27-item Intolerance of Uncertainty Scale (Freeston et al., 1994). Items are scored on a 5-point Likert scale ranging from 1 to 5.
Rejection sensitivity (C-RSQ; Downey et al., 2013) | Baseline, Month 2, 6, 9 and 12
  The "Children's Rejection Sensitivity Questionnaire" (C-RSQ; Downey et al., 1998) assesses the rejection sensitivity through 6 hypothetical interpersonal situations with ambiguous outcomes. Participants indicate on a 6-point Likert scale whether they would be nervous about the situation, how angry they would be about the situation, and what their outcome expectancy is.
Satisfaction with the intervention (ZUF-8; Schmidt et al., 1989) | Week 8
  The ZUF-8 is a questionnaire with 8 items for the global, one-dimensional assessment of patient satisfaction (Schmidt et al., 1989).
Adherence to the online-intervention | During the eight-week online-intervention
  Assessed within the online-intervention. Indicator of adherence: time spent in program.
Adherence | During the eight-week online-intervention
  Assessed within the online-intervention. Indicator of adherence: number of clicks.
Adherence | During the eight-week online-intervention
  Assessed within the online-intervention. Indicator of adherence: number of modules completed.
Adherence | During the eight-week online-intervention
  Assessed within the online-intervention. Indicator of adherence: number of exercises completed.
Negative Intervention Effects (INEP; Ladwig, Rief & Nestoriuc, 2014) | Week 8
  Negative effects of the intervention will be assessed using a version of the "Inventory for the Assessment of Negative Effects in Psychotherapy" (Kinder-INEP; Bieda et al., 2018; INEP; Ladwig et al., 2014) adapted for online interventions and for children and adolescents. 12 Items.
Working Alliance (WAI-CA; Figueiredo, 2016) | Week 2, 4, 6, 8
  The "Working Alliance Inventory for guided Internet Interventions" (WAI-I; Gómez Penedo et al., 2020) is a self-report questionnaire that measures therapeutic alliance in online interventions with therapeutic support. "Working Alliance Inventory for Children and Adolescents" (WAI-CA) consists of 12 items and has good psychometric properties (Gómez Penedo et al., 2020).
Therapy Motivation (MYTS; Breda & Riemer, 2012) | Baseline, Week 2, 4, 6, 8
  The "Motivation for Youth's Treatment Scale" (MYTS; Breda & Riemer, 2012) measures youth's motivation for therapy through a self-report questionnaire. The MYTS is a psychometrically based scale consisting of 8 items. Responses are rated on a 5-point likert scale. Higher ratings indicate higher motivation.
Acute suicidality | Baseline, Month 12
  Assessed by the Kinder-DIPS interview (Margraf et al., 2017; Schneider et al., 2017).
Acute suicidality | Baseline, Week 2, 4, 6, Month 2, 6, 9, 12
  Suicidality will throughout the study be evaluated by the item 9 of the "Patient Health Questionnaire-9 for Adolescents" (i.e., PHQ-A; Johnson et al., 2002). With a score "3" as the highest score.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie J Schmidt, Prof. Dr., Principal Investigator — University of Bern, Devision of Clinical Child and Adolescent Psychology
Locations (1):
- University of Bern, Division of Clinical Child and Adolescent Psychology, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hirsig A, Hafeli XA, Schmidt SJ. Efficacy of a transdiagnostic Internet prevention approach in adolescents (EMPATIA study): study protocol of a randomized controlled trial. Trials. 2024 Aug 8;25(1):530. doi: 10.1186/s13063-024-08241-3. PMID 39118136
- See also: Homepage with study information for adolescents and care giver/parents — https://selfhelp.psy.unibe.ch/empatia/homepage